CLINICAL TRIAL: NCT07170813
Title: The Effect of Different Hyperextension Braces on Spinal Mobility
Brief Title: Effects of Different Hyperextension Braces on Spinal Mobility
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Tahsin Ozer (Other)
Responsible Party: Sponsor-Investigator, Mustafa Tahsin Ozer, Research assisstant, Izmir University of Economics
Organization: Izmir University of Economics (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2024/4; Yalova University (Other: Yalova University Scientific Research Project)
Record Dates: First submitted 2025-08-11; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Corset; Spinal Mobility; Posture
Keywords: Posture; movement; biomechanics; corset; spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinomed (Experimental): In this study, the effects of the Spinomed brace on spinal mobility will be evaluated. Participants will be fitted with the Spinomed brace for a defined period, and spinal range of motion will subsequently be assessed. Measurements will be performed using the dual inclinometer method, which provides an objective and reliable evaluation of spinal movements, including flexion, extension, lateral flexion, and rotation. The data obtained will be analyzed to determine the impact of the Spinomed brace on spinal mobility and to contribute to evidence-based clinical practice.
  Interventions: Other: Spinal hyperextension brace
- Jewett (Experimental): In this study, the effects of the Jewett brace on spinal mobility will be evaluated. Participants will be fitted with the Jewett brace for a defined period, and spinal range of motion will subsequently be assessed. Measurements will be performed using the dual inclinometer method, which provides an objective and reliable evaluation of spinal movements, including flexion, extension, lateral flexion, and rotation. The data obtained will be analyzed to determine the impact of the Jewett brace on spinal mobility and to contribute to evidence-based clinical practice.
  Interventions: Other: Spinal hyperextension brace

INTERVENTIONS:
Other: Spinal hyperextension brace — The Jewett brace is a hyperextension spinal orthosis designed to limit spinal flexion and promote proper posture by applying anterior and posterior forces to the thoracolumbar spine. It is commonly used for spinal fractures, postural disorders, and to reduce spinal load. Participants will wear the Jewett brace during the intervention phase, and spinal mobility and posture will be assessed.

SUMMARY:
This project aims to investigate the effects of different hyperextension braces (Jewett and Spinomed) on spinal mobility and posture. Hyperextension braces are commonly prescribed to limit spinal flexion and regulate load distribution, especially in cases of spinal injuries and postural disorders. However, their objective impact on spinal biomechanics remains unclear.

Purpose and Scope The study will be conducted on 30 healthy participants aged 18-35.

Spinal mobility, posture, and movement analysis will be assessed using a dual inclinometer and the PostureScreen mobile application.

Evaluations will be performed under three conditions:

* Without a brace
* With a Jewett brace
* With a Spinomed brace (applied in randomized order)

Assessments will include four-direction spinal mobility and postural analysis during daily life activities such as standing, squatting, and single-leg stance.

Hypotheses H0: Hyperextension braces do not restrict spinal mobility. H1: Hyperextension braces restrict spinal mobility. H2: Hyperextension braces do not alter body alignment during movements. H3: Hyperextension braces alter body alignment during movements.

Methodology

The study is designed as a cross-sectional trial.

Each measurement will be repeated three times. Data will be analyzed statistically using ANOVA or Kruskal-Wallis tests depending on distribution.

Ethical approval has been obtained (Yalova University, Protocol No: 2024/4).

Expected Contributions Academic: Results are expected to be presented at the Congress of the International Society of Biomechanics (2025) and published in a high-impact Q1 journal such as Spine.

Clinical: Findings will provide objective data on the effectiveness of hyperextension braces, guiding clinicians and physiotherapists in brace selection.

Educational: The project will also contribute to the training of young researchers, offering hands-on experience in research design and execution

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged 18-35.
* Body mass index (BMI) between 18.5 and 24.9 kg/m2

Exclusion Criteria:

* Having experienced pain, discomfort, or discomfort in the upper back, waist, or lower extremities in the last 4 weeks on the Nordic Musculoskeletal System Questionnaire.
* A score above 20 on the Oswestry Disability Questionnaire.
* Having a condition related to spinal malalignment identified by a specialist physician (such as scoliosis, hyperkyphosis, hypokyphosis, Schuerman's kyphosis).
* Having a history of congenital hip dislocation.
* Having had surgery on the lower extremities or spine.
* Having a neurological disease or medication use that could cause balance loss.
* Having engaged in regular exercise in the last 6 months.
* Having a history of regular brace use in the last 6 months.
* Having a rheumatic disease affecting the axial skeleton.
* Having a diagnosis of a disease related to the axial skeleton, such as spondylosis, spondylolisthesis, spinal stenosis, or disc herniation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Spinal Mobility (Range of Motion) | 11 months
  Sppinal ROM in flexion, extension, and lateral flexions will be measured using dual inclinometers to assess the impact of each brace.

SECONDARY OUTCOMES:
Postural Alignment Scores via PostureScreen App | 11 months
  Postural alignment will be assessed using the PostureScreen mobile application. Key parameters such as head shift, shoulder asymmetry, and thoracic kyphosis will be recorded to evaluate the impact of each brace condition.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep İclal Sag, Study Director — University of Yalova
Locations (1):
- University of Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No